CLINICAL TRIAL: NCT06578117
Title: Statistical Learning as a Novel Intervention for Cortical Blindness
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Matthew Cavanaugh, Research Assistant Professor, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00009495
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Stroke, Ischemic; Hemianopia, Homonymous; Hemianopsia; Occipital Lobe Infarct; Visual Field Defect, Peripheral; Vision Loss Partial; Quadrantanopia; Stroke Hemorrhagic
Keywords: occipital stroke; vision loss after stroke; vision recovery; vision restoration; partial vision loss
MeSH Terms: conditions — Ischemic Stroke; Hemianopsia; Hemorrhagic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Visual Training in Cortically Blind cohort (Experimental)
  Interventions: Device: Vision Training and Learning Task
- Visual Training in Control cohort (Experimental)
  Interventions: Device: Vision Training and Learning Task

INTERVENTIONS:
Device: Vision Training and Learning Task — Participants will be seated at a computer, and will be shown a random-noise visual stimulus drifting in one of eight directions. Participants will be instructed to indicate the direction of motion they perceive using a Sony Access Controller or a computer keyboard. Sound cues during stimulus presentation will also be used to ensure participants are aware of stimulus onset during the training task.
  After several repetitions of this visual training, a second set of visual cues will be presented to evaluate participant's learning of the program. Responses will be provided in the same manner by input from the controller or the keyboard.

SUMMARY:
This project aims to develop a novel visual training paradigm for use in visually-intact participants and those sufferings from stroke-induced visual impairments. Our task design is built upon theories of statistical learning to reduce the overall training burden while still producing profound improvements to visual abilities. Efficacy will be first established in visually-intact controls before testing in stroke survivors to assess the feasibility of this form of learning in the damaged visual system.

ELIGIBILITY:
Cortically Blind participants

Inclusion criteria:

* Between 21 and 75 years of age
* Residents of the United States or Canada
* Have successfully completed previous enrollment in Dr. Huxlin study (IRB #5966 or #75)
* Exhibit unilateral stroke or stroke-like damage to primary visual cortex or its immediate afferent white matter sustained within the specified age range of 21 - 75 years (verified by MRI and/or CT scans)
* Reliable visual field defects in both eyes (homonymous defects) as measured by Humphrey visual fields. This deficit must be large enough to enclose a 5-deg diameter visual stimulus.
* Able to fixate on visual targets reliably for 1000ms within 1-deg of visual angle.
* Willing, able, and competent to provide their own informed consent
* Normal cognitive abilities and be able to understand written and oral instructions in English

Exclusion criteria:

* Past or present ocular disease interfering with visual acuity
* Best corrected visual acuity (BCVA) worse than 20/40 in either eye
* Sustained documented or suspected damage to the dorsal Lateral Geniculate Nucleus
* Presence of diffuse whole brain degenerative processes
* History of traumatic brain injury
* Any other brain damage deemed by study staff to potentially interfere with training ability or outcome measures
* Documented history of drug/alcohol abuse
* Currently taking neuroactive medications which would impact training, as determined by PI
* Cognitive or seizure disorders
* One-sided attentional neglect
* Those who lack the competence or are otherwise unable to perform the visual training exercises as directed.

Control participants

Inclusion criteria:

* Between 21 and 75 years of age
* No history of neurological disorder.
* Competent and responsible, as determined by the screening interview

Exclusion criteria:

* Any damage to the visual system
* Those who are suffering from an active disease process involving their nervous system.
* Presence of cognitive or seizure disorders
* Best corrected visual acuity worse than 20/40 in either eye
* Presence of visual field loss from ocular disease or disorder

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Explicit Learning - Response Time | Baseline
  Reaction time (ms) when performing motion discriminations for the final stimulus of a statistically-linked triplet will be compared against reaction times for stimuli with identical motion directions, presented with alternative placement within a triplet. Comparisons will be made only for correct responses in the final 20% of overall testing session trials.
Implicit Learning - Triplet Familiarity | Baseline
  Participant familiarity with statistically-linked triplets of motion will be assessed via a two-interval, forced-choice task. Familiarity will be measured as a percentage of comparisons in which the more prevalent triplet is selected as more familiar. Familiarity of high-probability, low-probability, and null-probability triplets will be compared following training.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No